CLINICAL TRIAL: NCT03936309
Title: A Comparison of Scar Infiltration, Scar Deactivation, and Standard of Care for the Treatment of Chronic, Post-Surgical Pain After Cesarean Section in the Primary Care Setting: A Comparative Effectiveness Trial.
Brief Title: A Comparison of Scar Infiltration, Scar Deactivation, and Standard of Care for the Treatment of Chronic, Post-Surgical Pain After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Loomis (U.S. Federal Agency)
Collaborators: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jennifer Loomis, Principal Investigator, 375th Medical Group, Scott Air Force Base
Organization: 375th Medical Group, Scott Air Force Base (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20190005H
Record Dates: First submitted 2019-04-25; First posted 2019-05-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Scar; Cesarean Section; Dehiscence
MeSH Terms: conditions — Cicatrix | interventions — Lidocaine; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scar Deactivation Surface Release (Experimental): Alternating placement of Spring Ten (0.30x40 mm) acupuncture needles to surround scar left in place for a treatment duration of 20 minutes. Needles will be placed at intervals of 1cm to 1.5 cm and will surround the scar with a maximum of 20 needles per treatment.
  Interventions: Other: Scar Deactivation Surface Release Technique protocol
- Scar Infiltration with 0.25-1% Lidocaine (Experimental): Will consist of calculation of 3 mg/kg dose of 0.5-1% Lidocaine and a dermal followed by subcutaneous injection using 1.5 inch 25 G needle and syringe appropriate for volume based on calculated dose.
  Interventions: Other: Scar Infiltration with 0.25-1% Lidocaine
- Physical Therapy (Experimental): Will be a referral to physical therapy specifying McKenzie protocol treatment for the presenting complaint. The McKenzie protocol is a form of standard of care physical therapy in which the physical therapist tries to find a cause and effect relationship between the positions the patient usually assumes while sitting, standing, or moving, and the location of pain because of those positions or activities. The therapeutic approach requires a patient to move through a series of activities and test movement to gauge the patient's pain response. The approach then uses that information to develop an exercise program designed to centralize or alleviate the pain.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Scar Deactivation Surface Release Technique protocol — ▪ Alternating placement of Spring Ten (0.30x40 mm) acupuncture needles to surround scar left in place for a treatment duration of 20 minutes. Needles will be placed at intervals of 1cm to 1.5 cm and will surround the scar with a maximum of 20 needles per treatment.
  Arms: Scar Deactivation Surface Release
Other: Scar Infiltration with 0.25-1% Lidocaine — ▪ Will consist of calculation of 3 mg/kg dose of 0.5-1% Lidocaine and a dermal followed by subcutaneous injection using 1.5 inch 25 G needle and syringe appropriate for volume based on calculated dose.
  Arms: Scar Infiltration with 0.25-1% Lidocaine
Other: Physical therapy — ▪ Will be a referral to physical therapy specifying McKenzie protocol treatment for the presenting complaint. The McKenzie protocol is a form of standard of care physical therapy in which the physical therapist tries to find a cause and effect relationship between the positions the patient usually assumes while sitting, standing, or moving, and the location of pain because of those positions or activities. The therapeutic approach requires a patient to move through a series of activities and test movement to gauge the patient's pain response. The approach then uses that information to develop an exercise program designed to centralize or alleviate the pain.
  Arms: Physical Therapy

SUMMARY:
To compare scar infiltration with 0.5-1% Lidocaine at a dose of 3 mg/kg (max dose 300 mg) or scar deactivation with acupuncture surface release technique to determine which is more effective in reducing pain in adult patients with chronic, post-surgical pain related to the site of incision after low transverse Cesarean section compared to standard of care physical therapy with the McKenzie Method.

DETAILED DESCRIPTION:
While there is not a clearly established and widely accepted pathophysiological cause to this post-operative pain, studies have estimated that between 7-33% of patients experience chronic peri-incisional pain after Cesarean section with Pfannenstiel incision - a type of abdominal surgical incision that allows access to the abdomen and the most common method for performing Cesarean sections today - defined as pain persisting beyond the period of expected healing, approximately 3 months.

Management of chronic peri-incisional pain after Cesarean section requires an extensive workup including laboratory testing (CBC, ESR, Urinalysis, STI testing) and imaging (transvaginal ultrasonography and abdominal CT) to rule out organic causes. Once a visceral etiology from postoperative pain has been excluded, there is not a well-established guideline dictating standard of care, however treatment can include analgesics such as Acetaminophen or Non-Steroidal Anti-inflammatory Drugs, and in refractory cases suggestive of neuropathic pain Tricyclic Antidepressants, Gabapentin, Pregabalin, and Serotonin-Norepinephrine Reuptake Inhibitors can be used. If medicinal therapy fails to manage symptoms, consultation for pain management specialists and/or surgical evaluation is often considered.

Scar deactivation is used as standard of care for treatment and resolution of scar associated pain in patients with a history of Cesarean section by medical acupuncturists, both abdominal and/or low back pain that began after the cesarean section. Scar infiltration with lidocaine has been used in numerous clinical settings, masquerading under different names. Referred to as Neural Therapy in Germany, the technique of injecting short-acting local anesthetic into the dermal subcutaneous junction of scar tissue has been widely applied; however there is limited readily available clinical trial evidence supporting its reported effectiveness. Theoretically, it is postulated that the anti-inflammatory effects of local anesthetics play a role in mitigating the autonomic nervous system disruption of interference fields caused by scar tissue. Local anesthetics promote anti-inflammatory activity through a variety of mechanisms including reversibly inhibiting leukocyte adhesion by interfering with the action of integrins and leukocyte adhesion molecule-1, limiting leukocyte migration, reversible inhibition of phagocytosis, inhibition of phospholipase A2, inhibition of prostaglandins, inhibition of thromboxane release, inhibition of leukotriene release, inhibition of histamine release, reduction in free radical formation, and inhibition of cytokine release. Additionally, Lidocaine injection is proposed to alleviate nerve entrapment within fascia through hydrodissection, a technique being effectively utilized in the management of carpal tunnel syndrome.

Scar deactivation is the technique of inserting acupuncture needles at a 30-45 degree angle into the superficial fascia to surround a scar. It is postulated that needle insertion into connective tissue produces analgesia through a multifaceted process encompassing the disruption and remodeling of extracellular matrix in loose connective tissue, alterations in gene expression affecting neurotransmitter levels, and cellular signaling pathways impacted in response to fibroblast and mast-cell involvement. In traditional Chinese medicine, injuries resulting in scar tissue formation are thought of as areas of blood and subsequently Qi stagnation. Disruptions in the flow of Qi at the point of scar tissue can result in abnormal skin sensations such as pain, itching, and numbness in addition to systemic effects. A case report has demonstrated effective pain relief in with an acupuncture protocol utilizing scar deactivation technique.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base or Scott AFB (a military installation) in order to participate in this study.**

Inclusion Criteria:

* Female DoD beneficiaries age 18 years or older
* 3 months or greater postpartum with abdominal and/or back pain starting after low transverse Cesarean section scar.
* If subject has had prior Scar Deactivation with Surface Release Technique for cesarean section scar they must have completed a washout period of 12 weeks or more.

Exclusion Criteria:

* Pregnant
* Prior Scar Deactivation with Surface Release Technique for cesarean section scar within the last 12 weeks.
* Ever had Prior Scar Infiltration with Lidocaine for cesarean section.
* Active cellulitis surrounding scar
* Revision of Cesarean section scar
* Vertical incision or emergent Cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Change in Defense and Veterans Pain Rating Scale (DVPRS) between each time frame | time 0, 4 weeks, 8 weeks, 16 weeks, 20 weeks
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
  The goal for pain reductions will be 50% as a primary outcome.
Change in Patient and Observer Scar Assessment Scale (POSAS) between each time frame | time 0, 4 weeks, 8 weeks, 16 weeks, 20 weeks
  The Patient and Observer Scar Assessment Scale consists of the total score of two numeric scales measured by the patient and a qualified observer. Each scale assesses the scar by six characteristics on 10-point scales with a 1 corresponding to normal skin and a 10 representing the worst imaginable condition for that characteristic. The Total Score of both scales is calculated by summing scores of the six items resulting in a range of 6 to 60. The POSAS is treated as an interval variable; therefore, parametric methods will be used for this outcome.

SECONDARY OUTCOMES:
Single question asking if subjects' expectations were met? -- Binary yes/no | 20 weeeks
  Ask if the subjects' expectations were met regarding physical therapies/lidocaine/acupuncture effectiveness for chronic, post-surgical pain related to low transverse Cesarean Section. Answer is Yes/No.
Single question asking subjects' change in pain severity reported as a percentile (10%, 20%, ...) | 20 weeks
  Report as a percentage, where the greater the percent the greater the pain reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- 375th Medical Group, Scott Air Force Base, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJ, Driscoll AK, Mathews TJ. Births: Final Data for 2015. Natl Vital Stat Rep. 2017 Jan;66(1):1. PMID 28135188
- [Background] Wasserman JB, Steele-Thornborrow JL, Yuen JS, Halkiotis M, Riggins EM. Chronic caesarian section scar pain treated with fascial scar release techniques: A case series. J Bodyw Mov Ther. 2016 Oct;20(4):906-913. doi: 10.1016/j.jbmt.2016.02.011. Epub 2016 Mar 10. PMID 27814873
- [Background] Okabayashi K, Ashrafian H, Zacharakis E, Hasegawa H, Kitagawa Y, Athanasiou T, Darzi A. Adhesions after abdominal surgery: a systematic review of the incidence, distribution and severity. Surg Today. 2014 Mar;44(3):405-20. doi: 10.1007/s00595-013-0591-8. Epub 2013 May 9. PMID 23657643
- [Background] Suleiman S, Johnston DE. The abdominal wall: an overlooked source of pain. Am Fam Physician. 2001 Aug 1;64(3):431-8. PMID 11515832
- [Background] Srinivasan R, Greenbaum DS. Chronic abdominal wall pain: a frequently overlooked problem. Practical approach to diagnosis and management. Am J Gastroenterol. 2002 Apr;97(4):824-30. doi: 10.1111/j.1572-0241.2002.05662.x. PMID 12003414
- [Background] Loos MJ, Scheltinga MR, Mulders LG, Roumen RM. The Pfannenstiel incision as a source of chronic pain. Obstet Gynecol. 2008 Apr;111(4):839-46. doi: 10.1097/AOG.0b013e31816a4efa. PMID 18378742
- [Background] Speer LM, Mushkbar S, Erbele T. Chronic Pelvic Pain in Women. Am Fam Physician. 2016 Mar 1;93(5):380-7. PMID 26926975
- [Background] Brobyn TL, MK Chung, and PJ LaRiccia "Neural therapy: An overlooked game changer for patients suffering chronic pain?" J Pain Relief 2015;4: 184.
- [Background] Weinschenk S. "Neural therapy--A review of the therapeutic use of local anesthetics" Acupuncture and Related Therapies 2012.
- [Background] Egli S, Pfister M, Ludin SM, Puente de la Vega K, Busato A, Fischer L. Long-term results of therapeutic local anesthesia (neural therapy) in 280 referred refractory chronic pain patients. BMC Complement Altern Med. 2015 Jun 27;15:200. doi: 10.1186/s12906-015-0735-z. PMID 26115657
- [Background] Hollmann MW, Durieux ME. Local anesthetics and the inflammatory response: a new therapeutic indication? Anesthesiology. 2000 Sep;93(3):858-75. doi: 10.1097/00000542-200009000-00038. No abstract available. PMID 10969322
- [Background] Cassuto J, Sinclair R, Bonderovic M. Anti-inflammatory properties of local anesthetics and their present and potential clinical implications. Acta Anaesthesiol Scand. 2006 Mar;50(3):265-82. doi: 10.1111/j.1399-6576.2006.00936.x. PMID 16480459
- [Background] Malone, D, T Clark, and N Wei. "Ultrasound-guided percutaneous injection, hydrodissection, and fenestration for carpal tunnel syndrome: description of a new technique." Journal of Applied Research. 2010;10(3):116-123.
- [Background] Liddle CE, Harris RE. Cellular Reorganization Plays a Vital Role in Acupuncture Analgesia. Med Acupunct. 2018 Feb 1;30(1):15-20. doi: 10.1089/acu.2017.1258. PMID 29410716
- [Background] Fang S. The successful treatment of pain associated with scar tissue using acupuncture. J Acupunct Meridian Stud. 2014 Oct;7(5):262-4. doi: 10.1016/j.jams.2014.05.001. Epub 2014 Jun 24. PMID 25441952

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03936309/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03936309/ICF_001.pdf